CLINICAL TRIAL: NCT02310230
Title: An Evaluation of the Utility of the ExSpiron Respiratory Variation Monitor During Upper GI Endoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Donald Mathews (Other)
Collaborators: Respiratory Motion, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Donald Mathews, Attending Anesthesiologist and Professor of Anesthesiology, University of Vermont
Organization: University of Vermont (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: M14-281
Record Dates: First submitted 2014-09-18; First posted 2014-12-08 (Estimated); Results first posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-05

CONDITIONS: Biliary Tract Diseases; Stomach Neoplasms; Carcinoma, Pancreatic Ductal; Barrett Esophagus
Keywords: Endoscopy, Upper; Minute Ventilation; Tidal Volume; Respiratory Rate
MeSH Terms: conditions — Biliary Tract Diseases; Stomach Neoplasms; Carcinoma, Pancreatic Ductal; Barrett Esophagus

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Blinded Group (Other): Data from the ExSpiron Respiratory Variation Monitor (minute ventilation, tidal volume, and respiratory rate) will not be displayed. The anesthesia provider will care for the patient in the usual manner.
  Interventions: Device: ExSpiron Respiratory Variation Monitor
- Monitor Group (Experimental): The ExSpiron Respiratory Variation Monitor will display continuous real-time measurements of minute ventilation, tidal volume, and respiratory rate, and the anesthesia provider will be instructed to utilize this information in the care of the patient as they deem appropriate.
  Interventions: Device: ExSpiron Respiratory Variation Monitor

INTERVENTIONS:
Device: ExSpiron Respiratory Variation Monitor — Non-invasive monitoring of minute ventilation, tidal volume, and respiratory rate.

SUMMARY:
Purpose: To assess the utility of a new medical device that monitors a patient's breathing during medical procedures in which a patient is sedated, but not mechanically ventilated. In minor procedures, such as endoscopy (where the doctor examines a patient's digestive tract by a TV camera inserted through the mouth), patients do not require general anesthesia, in which a machine would take over their breathing while they are unconscious for surgery. However, during endoscopic procedures it is sometimes difficult for the anesthesiologist to monitor the patient's breathing-specifically, to monitor changes in breathing patterns and the adequacy of breathing. In endoscopy procedures, the room is darkened, and the patient's mouth is generally occupied by the endoscope. While the anesthesiologist can listen to the patient's breathing sounds with a stethoscope, this type of monitoring can only be done periodically, and there is limited ability to gauge the adequacy of ventilation. This study will use the ExSpiron Respiratory Volume Monitor (RVM), which measures non-invasive minute ventilation (MV), tidal volume (TV) and respiratory rate (RR), in patients undergoing an endoscopic procedure to provide additional information regarding the effects of clinical interventions such as drug administrations or airway maneuvers on the patient's respiratory status.

For patients who give informed consent, study participation means that they will have a PadSet consisting of 3 electrodes applied to the chest. Another component, a nasal cannula (a thin clear plastic tube that goes under the nose) will give patients supplemental oxygen, and is standard of care for endoscopy at UVM Medical Center. Patients will then be asked to breathe in and out of a portable spirometer (breath meter) for 30 seconds up to five times. This data will be compared to data recorded by the monitor to confirm that the monitor is recording accurately. The procedure will then go forward in the normal fashion. Patients will be randomly placed into one of two groups. In the first group during the procedure, the anesthesiologist will not be able to see the numbers (MV, TV, and RR) displayed screen of the monitor, so the data will not be used to guide the patient's clinical care. In the second group, the anesthesiologist will be able to see the RVM measurements of MV, TV, and RR to evaluate the effect of the interventions. Monitoring for both groups will continue in the recovery room, until discharge.

DETAILED DESCRIPTION:
The purpose of this study is to assess the utility of the ExSpiron Respiratory Variation Monitor in patients undergoing an interventional procedure with anesthesia. The primary outcome measure will be the average minute ventilation of the patient during the procedure. This study will also examine the correlation between clinical interventions such as drug administrations or airway maneuvers with data from the monitor. Additionally the study may provide information about the ability of this new monitoring system to prevent hypoxemia during these procedures and to consider its utility, compared with capnography, to detect hypopnea.

Background Assessing the adequacy of ventilation during Monitored Anesthesia Care (MAC) and sedation is difficult. Agents used to provide procedural sedation can depress ventilatory drive and can interfere with airway patency, making it much more likely that the patient will hypoventilate and experience partial or complete obstruction to ventilation. [It is actually clinically easier to administer general anesthesia and insert an airway management device such as an endotracheal tube or a laryngeal mask airway , however given the superior recovery profile following sedation vs. general anesthesia, it is usually preferable to administer sedation, if the procedure can be performed with its use.] The American Society of Anesthesiologists maintains a database of closed malpractice claims which allows analysis of patterns of injury. A study considering claims from MAC/sedation cases found that 40% of the MAC claims resulted in death or brain damage, that 25% of the claims that were associated with oversedation/hypoventilation occurred in the endoscopy suite, and that 44% of the oversedation cases could have been prevented by better monitoring.1 A study comparing claims from remote locations (such as endoscopy) with operating rooms, found that 50% of remote location claims involving monitored anesthesia care, the proportion of claims for death was increased in remote location claims [54 vs. 29% (operating room claims)], respiratory damaging events were more common in remote location claims (44 vs. 20%), with inadequate oxygenation/ventilation the most common specific event (21 vs. 3% in operating room claims), and that remote location claims were more often judged as being preventable by better monitoring (32 vs. 8% for operating room claims).2

Upper endoscopy procedures, such as upper GI endoscopy and endoscopic retrograde cholangiopancreatography (ERCP), are particularly challenging where the anesthesiologist has limited access to the patient's head and is working in darkened rooms. Indeed investigators have found it very difficult to find a combination of propofol and short acting opioid that allows instrumentation of the esophagus without "intolerable ventilatory depression".3 Trying to assess ventilation by observing chest excursion or listening to ventilation with a stethoscope under these conditions can be difficult and can be done only periodically. Side-stream nasal cannula end-tidal capnography offers a possible solution, but the cannula can become dislodged and the proceduralist's endoscope often interferes with its function. End-tidal capnography in the non-intubated patient is very insensitive to changes in minute ventilation. At best, this technology can usually assess only the presence or absence of ventilation: there is limited ability to judge the adequacy of ventilation or to quantify it.4

The Study Device The ExSpiron Respiratory Volume Monitor (Respiratory Motion, Inc., Waltham MA) has FDA 501(k) clearance to be used for patient care. It consists of a proprietary PadSet that is placed on the chest in the mid-axillary line and connected to a free standing monitor. This monitor measures and analyzes the changes in thoracic electrical impedance that occur during the respiratory duty cycle. It is able to quantify respiratory rate and also determine tidal volume and minute ventilation as well as graphically display changes in lung volumes. It has been shown to accurately measure the effect of interventions (medications, airway maneuvers) in endoscopy patients.5 Preliminary work has determined optimal lead placement demonstrated excellent correlation to spirometry with an R value of 0.94-0.98 and excellent accuracy and precision.6

Preliminary work cited below has shown that the monitor provides information about the effect of medications and airway maneuvers on breathing patterns that is not available with routine monitoring. This study seeks to extend that knowledge by investigating whether using this information in real-time results in different respiratory measurements compared to patients with routine monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Subjects undergoing upper gastrointestinal endoscopy

Exclusion Criteria:

* Patients with a history of thoracotomy with resection of lung tissue
* Patients with a history of severe chronic obstructive pulmonary disease (defined as an inability to climb a flight of stairs or FEV1/VC of less than 30% of predicted)
* BMI greater than 43.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-09-22 (Actual); Primary Completion 2016-05-09 (Actual); Study Completion 2016-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald M Mathews, M.D., Principal Investigator — University of Vermont
Locations (1):
- University of Vermont Medical Center, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bhananker SM, Posner KL, Cheney FW, Caplan RA, Lee LA, Domino KB. Injury and liability associated with monitored anesthesia care: a closed claims analysis. Anesthesiology. 2006 Feb;104(2):228-34. doi: 10.1097/00000542-200602000-00005. PMID 16436839
- [Background] Metzner J, Posner KL, Domino KB. The risk and safety of anesthesia at remote locations: the US closed claims analysis. Curr Opin Anaesthesiol. 2009 Aug;22(4):502-8. doi: 10.1097/ACO.0b013e32832dba50. PMID 19506473
- [Background] LaPierre CD, Johnson KB, Randall BR, White JL, Egan TD. An exploration of remifentanil-propofol combinations that lead to a loss of response to esophageal instrumentation, a loss of responsiveness, and/or onset of intolerable ventilatory depression. Anesth Analg. 2011 Sep;113(3):490-9. doi: 10.1213/ANE.0b013e318210fc45. Epub 2011 Mar 17. PMID 21415430
- [Background] Holley K, Mathews D, Freeman J, Brayanov J, Schapiro H. The Use of a Respiratory Volume Monitor to Assess Ventilation Before & After Airway Maneuvers during Upper Endoscopy. Poster Presentation, American Society of Anesthesiologists, October 2013, San Francisco, CA
- [Background] Voscopoulos C, Brayanov J, Ladd D, Lalli M, Panasyuk A, Freeman J. Special article: evaluation of a novel noninvasive respiration monitor providing continuous measurement of minute ventilation in ambulatory subjects in a variety of clinical scenarios. Anesth Analg. 2013 Jul;117(1):91-100. doi: 10.1213/ANE.0b013e3182918098. Epub 2013 Jun 3. PMID 23733842
- [Background] Freeman J, Lalli M, Yocum N, Panasyuk A, Panasyuk S, and Lew R, 328: Non-invasive Monitoring of Tidal Volume and Minute Ventilation in Non-intubated Patients. Critical Care Medicine, 2011. 39(12): p. 88 10.1097/01.ccm.0000408627.24229.88.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Blinded Group | Monitor Group
Started | 50 | 50
Completed | 41 | 32
Not Completed | 9 | 18
Not completed — Physician Decision | 1 | 3
Not completed — monitor baseline taken after induction | 2 | 7
Not completed — Poor signal quality | 5 | 8
Not completed — Case cancelled | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Blinded Group | Monitor Group | Total
Number analyzed (Participants) | 41 | 32 | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.9 (17.0) | 60.5 (11.0) | 56.2 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 16 | 39
  Male | 18 | 16 | 34
Height [Mean (Standard Deviation); unit: centimeters] | 169.5 (9.7) | 169.3 (12.0) | 169.4 (10.8)
Weight [Mean (Standard Deviation); unit: kilograms] | 82.1 (23.8) | 75.3 (17.1) | 79.1 (21.4)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.3 (6.9) | 26.2 (5.0) | 27.4 (6.2)
Length of Procedure [Mean (Standard Deviation); unit: minutes] | 30.1 (1.9) | 37.2 (3.2) | 33.2 (1.8)
Intra-Op Propofol [Mean (Standard Deviation); unit: mcg/kg/min] | 239.7 (108.2) | 241.4 (112.6) | 240.4 (110.2)

OUTCOME MEASURES:

1. Primary Outcome: Average Minute Ventilation in Patients Cared for Using the ExSpiron Respiratory Variation Monitor (RVM) Compared to Patients With Routine Monitoring in Patients Undergoing Upper Gastrointestinal Endoscopy
Description: Minute ventilation (or respiratory minute volume) is defined as the volume of air that can be inhaled or exhaled during one minute. The ExSpiron Respiratory Variation Monitor is able to quantify respiratory rate and also determine tidal volume and minute ventilation. The monitor measures a patient's baseline minute ventilation (MV) at the beginning of the case, and then compares subsequent minute volumes to that baseline, measured as a percentage of the baseline. In that respect, the minute ventilation (MV) values can often exceed 100 percent.
Time Frame: Duration of procedure: Approximately 60 minutes
Measure: Mean (Standard Error); unit: % of minute ventilation baseline
Arm/Group | Blinded Group | Monitor Group
Number analyzed (Participants) | 41 | 32
% of minute ventilation baseline | 86.7 (5.9) | 109.8 (9.3)

2. Secondary Outcome: Incidence of Airway Maneuvers Required to Maintain Ventilation in Each Group
Time Frame: Duration of procedure: Approximately 60 minutes
Measure: Mean (Full Range); unit: one airway maneuver
Arm/Group | Blinded Group | Monitor Group
Number analyzed (Participants) | 41 | 32
one airway maneuver | 2.2 [0 to 7] | 2.3 [0 to 8]

3. Secondary Outcome: Time With Low Minute Ventilation
Description: Percentage of procedure time spent with Minute Ventilation less than 40% of the Minute Ventilation Baseline. Minute ventilation (or respiratory minute volume) is defined as the volume of air that can be inhaled or exhaled during one minute. The ExSpiron Respiratory Variation Monitor is able to quantify respiratory rate and also determine tidal volume and minute ventilation.
Time Frame: Duration of Procedure: Approximately 60 Minutes
Measure: Mean (Standard Error); unit: percentage of procedure duration
Arm/Group | Blinded Group | Monitor Group
Number analyzed (Participants) | 41 | 32
percentage of procedure duration | 15.3 (2.8) | 7.1 (1.4)

ADVERSE EVENTS:
Arm/Group | Blinded Group | Monitor Group
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No